CLINICAL TRIAL: NCT02685020
Title: A Randomized, Parallel-group, Placebo-controlled, Double-blind Phase 1 Study in Healthy HIV-uninfected Adults to Evaluate Safety/Tolerability and Immunogenicity of Different Vaccine Schedules With Ad26.Mos.HIV and Clade C gp140
Brief Title: Safety, Tolerability and Immunogenicity Study of Different Vaccine Schedules With Ad26.Mos.HIV and Clade C Glycoprotein (gp)140 in Healthy Human Immunodeficiency Virus (HIV)-Uninfected Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Vaccines & Prevention B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CR108068; VAC89220HPX1002 (Other: Janssen Vaccines & Prevention B.V.)
Record Dates: First submitted 2016-02-12; First posted 2016-02-18 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Healthy
Keywords: Healthy; Human Immunodeficiency Virus; adenovirus serotype 26; Ad26.Mos.HIV; Vaccine; Placebo; Glycoprotein; IPCAVD010
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (6):
- Group 1A (Experimental): Participants will receive Ad26.Mos.HIV vaccine at Week 0 and 12; followed by Ad26.Mos.HIV vaccine + Clade C glycoprotein 140 vaccine containing 250 microgram (mcg) of total protein mixed with adjuvant (aluminum phosphate) at Week 24 and 48.
  Interventions: Biological: Ad26.Mos.HIV; Biological: Clade C gp140
- Group 1B (Placebo Comparator): Participants will receive placebo at weeks 0, 12, 24 and 48.
  Interventions: Drug: Placebo
- Group 2A (Experimental): Participants will receive Ad26.Mos.HIV vaccine + Clade C glycoprotein 140 vaccine containing 250 mcg of total protein mixed with adjuvant (aluminum phosphate) at Week 0, 12 and 24.
  Interventions: Biological: Ad26.Mos.HIV; Biological: Clade C gp140
- Group 2B (Placebo Comparator): Participants will receive placebo at weeks 0, 12 and 24.
  Interventions: Drug: Placebo
- Group 3A (Experimental): Participants will receive Ad26.Mos.HIV vaccine at Week 0; followed by Ad26.Mos.HIV vaccine + Clade C glycoprotein 140 vaccine containing 250 mcg of total protein mixed with adjuvant (aluminum phosphate) at Week 8 and 24.
  Interventions: Biological: Ad26.Mos.HIV; Biological: Clade C gp140
- Group 3B (Placebo Comparator): Participants will receive placebo at weeks 0, 8 and 24.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Ad26.Mos.HIV — Recombinant replication-deficient Ad26 vectored vaccine and consists of 3 Ad26 vectors, one containing a mosaic insert of envelope (Env) sequence, and 2 vectors containing mosaic inserts of Gag and Pol sequences (Ad26.Mos.1.Env + Ad26.Mos1.Gag-Pol + Ad26.Mos2.Gag-Pol). Total dose is 5*10^10 viral particle per 0.5 milliliter (mL) injection administered intramuscularly.
  Arms: Group 1A; Group 2A; Group 3A
Biological: Clade C gp140 — The Clade C gp140 vaccine containing 250 mcg of total protein, mixed with aluminum phosphate adjuvant, per 0.5 mL injection administered intramuscularly.
  Arms: Group 1A; Group 2A; Group 3A
Drug: Placebo — Normal saline, 0.5 mL injection administered intramuscularly.
  Arms: Group 1B; Group 2B; Group 3B

SUMMARY:
The primary purpose of this study is to assess safety, tolerability of the different vaccine schedules (different regimen durations and different number of dose administrations) with Ad26.Mos.HIV and Clade C Glycoprotein (gp) 140 and to assess Envelope (Env)-binding Antibody (Ab) responses of the different vaccine schedules.

DETAILED DESCRIPTION:
This is a phase 1 single-center, randomized (the study drug is assigned by chance), parallel group (each group of participants will be treated at the same time), placebo-controlled (study in which the experimental treatment or procedure is compared to a pretend treatment with no drug in it to test if the drug has a real effect), and double-blind (neither physician nor participant knows the treatment that the participant receives) study. Participants will be randomized in to 3 groups and will receive study vaccines or placebo. Group 1 will have 4 vaccination time points during 48 weeks, Groups 2 and 3 will have 3 vaccination time points during 24 weeks. The study comprises a Screening Period (up to 4 weeks), a Vaccination Period (maximum 48 weeks), and a Follow-up Period (up to 72 weeks). Participants' safety will be monitored throughout the study. An optional Long-term Extension (LTE) phase (approximately 1 year after Week 72) will be performed for participants randomized to receive study vaccine, who have received all planned vaccinations and are negative for HIV infection at Week 72. The duration of the participation will be approximately 124 weeks for participants participating to the optional LTE phase.

ELIGIBILITY:
Inclusion Criteria:

* Each participant must sign an informed consent form (ICF) indicating that he or she understands the purpose of and procedures required for the study and is voluntarily willing to participate in the study
* Participant must be healthy on the basis of physical examination, medical history, electrocardiogram (ECG), and vital signs measurement performed at Screening
* Participants are negative for Human Immunodeficiency Virus (HIV) infection at Screening
* All female participants of childbearing potential must have a negative serum pregnancy test (beta human chorionic gonadotropin [beta hCG]) at the Screening visit, and a negative urine pregnancy test pre-dose on Day 1
* Participants are willing/able to adhere to the prohibitions and restrictions specified in the protocol and study procedures

Exclusion Criteria:

* Participant has chronic hepatitis B or active hepatitis C, active syphilis infection, chlamydia, gonorrhea, or trichomonas . Active syphilis documented by serology unless positive serology is due to past treated infection
* In the 12 months prior to randomization, participant has a history of newly acquired herpes simplex virus type 2, syphilis, gonorrhea, non-gonococcal urethritis, chlamydia, pelvic inflammatory disease, trichomonas, mucopurulent cervicitis, epididymitis, proctitis, lymphogranuloma venereum, chancroid, or hepatitis B
* Participant has any condition for which, in the opinion of the investigator, participation would not be in the best interest of the participant (example, compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments
* Participant has had major surgery within 4 weeks prior to Screening or planned major surgery through the course of the study
* Participant has had a thyroidectomy or active thyroid disease requiring medication during the last 12 months

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2016-03-28 (Actual); Primary Completion 2018-01-05 (Actual); Study Completion 2019-01-03 (Actual)

PRIMARY OUTCOMES:
Titer to HIV-Envelope Specific Binding Antibodies Assessed by Env-Ab-binding Assay | Up to Week 72
Breadth of HIV-Envelope Specific Binding Antibodies Assessed by Env-Ab-binding Assay | Up to Week 72
Number of Participants With Local and Systemic Reactogenicity for 8 Days After Each Vaccination | Up to 8 days after each vaccination
  Participants will be asked to note occurrences of local reactions: pain/tenderness, erythema or swelling/induration at the injection site, and systemic events: fever (temperature measurement), fatigue, headache, nausea, myalgia and chills daily for 8 days post-vaccination. These occurrences will be recorded through the diary card provided to serve as a reminder to the participants for the next clinic visit.
Treatment Emergent Adverse Events (AEs) | Up to Week 72
Serious Adverse Events (SAEs) and AEs of Special Interest (AESI) | Up to Week 124
Discontinuations From Vaccination or From Study due to AEs | At the time of discontinuation from vaccination or from study (Up to Week 72)
Number of Participants With AEs or SAEs | Up to 28 days after each vaccination

SECONDARY OUTCOMES:
Env-Specific Functional Antibodies: Phagocytosis Score | Up to Week 72
Env-Specific Functional Antibodies: Breadths | Up to Week 72
Env-Specific Binding Antibody Isotypes: Titers | Up to Week 72
  The Isotyping (Clade C) (IgA, IgG1-4)- Env binding antibody titers will be assessed using ELISA.
Env-Specific Binding Antibody Isotypes: Breadths | Up to Week 72
  The Isotyping (Clade C) (IgA, IgG1-4)- Env binding antibody breadths will be assessed using ELISA.
Env-Specific Neutralizing Antibodies (nAbs): Titers | Up to Week 72
Env-Specific Neutralizing Antibodies (nAbs): Breadths | Up to Week 72
Induction of New T-cell Immune Response by the Vaccine | Up to Week 72
  Induction of new T-cell immune response against one or more of the vaccine epitopes using Interferon gamma Enzyme Linked Immuno spot assay (IFNg-ELISPOT assay) measuring Spot forming Units per 1 million peripheral blood mononuclear cells (SFU/1 mio PBMCs) above threshold (> 50 sfu/mio PBMC).
Change From Baseline of the Frequency of HIV-Specific PBMC and/or CD4 and/or CD8 T cells as Measured by ELISpot Interferon (IFN) Gamma | Up to Week 72

OTHER OUTCOMES:
Mucosal Immunogenicity | Up to week 72
  Immune Responses to the Different Vaccine Schedules in Mucosal Secretions.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Vaccines & Prevention B.V. Clinical Trial, Study Director — Janssen Vaccines & Prevention B.V.
Locations (1):
- Boston, Massachusetts, United States

REFERENCES:
- [Derived] Stephenson KE, Wegmann F, Tomaka F, Walsh SR, Tan CS, Lavreys L, Ansel JL, Kanjilal DG, Jaegle K, Nkolola JP, Peter L, Fogel R, Bradshaw C, Tyler A, Makoni T, Howe L, Quijada D, Chandrashekar A, Bondzie EA, Borducchi EN, Yanosick KE, Hendriks J, Nijs S, Truyers C, Tolboom J, Zahn RC, Seaman MS, Alter G, Stieh DJ, Pau MG, Schuitemaker H, Barouch DH. Comparison of shortened mosaic HIV-1 vaccine schedules: a randomised, double-blind, placebo-controlled phase 1 trial (IPCAVD010/HPX1002) and a preclinical study in rhesus monkeys (NHP 17-22). Lancet HIV. 2020 Jun;7(6):e410-e421. doi: 10.1016/S2352-3018(20)30001-1. Epub 2020 Feb 17. PMID 32078815